CLINICAL TRIAL: NCT05763121
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Assess the Efficacy, Safety, and Tolerability of Dexpramipexole Administered Orally for 52 Weeks in Participants With Severe Eosinophilic Asthma
Brief Title: A Study to Assess the Effect of Dexpramipexole in Adolescents and Adults With Severe Eosinophilic Asthma.
Acronym: EXHALE-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Program stopped due to the benefit risk profile no longer supports further development in the intended patient population.
Sponsor: Areteia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR-DEX-22-01; 2022-003004-33 (EudraCT Number); 2023049491 (Registry Identifier: Colombia CTA)
Record Dates: First submitted 2023-02-20; First posted 2023-03-10 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Eosinophilic Asthma; Asthma; Eosinophilic; Asthma
Keywords: Exacerbations; Severe Asthma; Dexpramipexole; EXHALE; Areteia; EXHALE-2; Uncontrolled Asthma; Asthma Attack
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 150 mg BID (Experimental): Dexpramipexole 150 mg oral tablet taken twice a day
  Interventions: Drug: Dexpramipexole Dihydrochloride
- 75 mg BID (Experimental): Dexpramipexole 75 mg oral tablet taken twice a day
  Interventions: Drug: Dexpramipexole Dihydrochloride
- Placebo (Placebo Comparator): Placebo oral tablet taken twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexpramipexole Dihydrochloride — oral administration of dexpramipexole tablet
  Arms: 150 mg BID; 75 mg BID
Drug: Placebo — oral administration of placebo tablet
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety of dexpramipexole as an adjunctive oral therapy in participants with inadequately controlled asthma with an eosinophilic phenotype and a history of asthma exacerbations.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo controlled, parallel group study designed to evaluate the efficacy and safety of dexpramipexole in adults and adolescents with severe, inadequately controlled asthma with eosinophilic phenotype on medium to high-dose inhaled corticosteroids (ICS )and at least one additional asthma controller medication with or without oral corticosteroids (OCS). Approximately 1400 participants will be randomized globally. Participants will receive dexpramipexole, or placebo, administered orally, over a 52-week treatment period. The study also includes a post-treatment follow-up period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form and assent form, as appropriate
2. Male or female ≥12 years of age at Screening Visit 1

   Asthma-related criteria
3. Documented physician diagnosis of asthma for ≥12 months prior to Screening Visit 1.
4. Treatment of asthma, participants must satisfy all the below (items a to c):

   1. Participants who have received asthma controller medication with medium or high dose inhaled corticosteroids (ICS; ≥500 μg/day fluticasone propionate dry powder formulation daily or clinically comparable, per Global Initiative for Asthma (GINA) 2021) on a regular basis for at least 12 months prior to Screening Visit 1.
   2. Documented treatment with a stable dose of either medium or high dose ICS for at least 3 months prior to Screening Visit 1. The ICS may be contained within an ICS/LABA (long-acting β2 agonist) combination product. Daily oral corticosteroids are an allowed concomitant medication; participants on daily oral corticosteroids must be on a stable dose for 3 months before Screening Visit 1.
   3. Use of one of more additional daily maintenance asthma controller medications according to standard practice of care is required. Use of a stable dose of any additional asthma controller medications must be documented for at least 3 months prior to Screening Visit 1.
5. Pre-bronchodilator forced expiratory volume (Pre-BD FEV₁) ≥40% and <80% (<90% for participants 12 to 17 years of age) of predicted at Screening Visit 2.
6. Variable airflow obstruction documented with at least one of the following criteria:

   1. Bronchodilator reversibility at Screening Visit 2, as evidenced by ≥12% and ≥200 mL improvement in FEV₁, 15 to 30 minutes following inhalation of 400 μg (four puffs) of albuterol/salbutamol (≥12% and ≥160 mL for ages 12 to17). Participants who do not meet the bronchodilator reversibility inclusion criterion but have ≥10% and ≥160 mL reversibility, may repeat the reversibility spirometry assessment once during the Screening period, at an unscheduled visit at least 7 days prior to baseline.
   2. Bronchodilator reversibility, using the criteria above, documented in the past 24 months prior to Screening Visit 1.
   3. Peak flow variation of ≥20% over a 2-week period, documented in the past 24 months prior to Screening Visit 1.
   4. Airflow variability in clinic FEV₁ ≥20% between two consecutive clinic visits, documented in the past 24 months prior to Screening Visit 1.
   5. Airway hyperresponsiveness (provocative concentration causing a 20% fall in FEV₁ of methacholine <8 mg/mL) documented in the past past 24 months prior to Screening Visit 1.
7. ACQ-6 ≥1.5 at Screening Visit 2.
8. Documented history of at least two asthma exacerbations requiring treatment with systemic corticosteroids (intramuscular, intravenous, or oral) within the past 12-month period prior to Screening Visit 1.

   General medical history
9. Negative urine pregnancy test for women of childbearing potential (WOCBP; after menarche) at the Screening Visit 2 and Baseline Visit.
10. WOCBP must use either of the following methods of birth control, from Screening Visit 1 through the End of Study Visit:

    1. A highly effective form of birth control (confirmed by the investigator). Highly effective forms of birth control include: true sexual abstinence, a vasectomized sexual partner, Implanon, female sterilization by tubal occlusion, any effective Intrauterine device (IUD), IUD/intrauterine system (IUS), Levonorgestrel Intrauterine system, or oral contraceptive.

       Or
    2. Two protocol acceptable methods of contraception in tandem.

       Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for ≥12 months prior to the planned date of the Baseline Visit without an alternative medical cause. The following age specific requirements apply:
    3. Women <50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone levels in the postmenopausal range.
    4. Women ≥50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.

Exclusion Criteria:

Asthma-related criteria

1. A participant who experiences a severe asthma exacerbation (defined as a deterioration of asthma that results in emergency treatment, hospitalization due to asthma, or treatment with systemic corticosteroids) at any time from 4 weeks prior to Screening Visit.

   Participants who experience an asthma exacerbation during the Screening/Run-in Period may remain in screening and proceed with study visits 14 days after they have completed their course of oral steroids or returned to their pre-Screening Visit maintenance dose of oral steroids and the investigator considers participant has returned to baseline status.
2. Current diagnosis of diseases which may confound interpretation of this study's findings such as allergic bronchopulmonary aspergillosis, eosinophilic granulomatosis with polyangiitis, eosinophilic gastrointestinal diseases, hypereosinophilic syndrome, chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis.
3. Respiratory infection: Upper or lower respiratory tract, sinus, or middle ear infection within the 4 weeks before Screening Visit 1.
4. For participants aged 12 to 17 years old, AEC of <0.15x10⁹/L at Screening Visit 1.

   Prohibited medications/procedures
5. Treatment with a biologic investigational drug in the last 5 months prior to Screening Visit 1. Treatment with non-biologic investigational drugs in the previous 30 days or five-half-lives prior to Screening Visit 1, whichever is longer. Treatment with GSK3511294 (long-acting anti-IL-5) in the past 12 months.
6. Treatment with any of the following monoclonal antibody therapies within 120 days prior to Baseline Visit: benralizumab, dupilumab, mepolizumab, reslizumab, omalizumab, tezepelumab, or tralokinumab.
7. Treatment with pramipexole (Mirapex®) within 30 days of Baseline Visit.
8. Treatment with selected drugs known to have a substantial risk of neutropenia in the past 30 days prior to Screening Visit 1.
9. Bronchial thermoplasty procedure in the past 12 months prior to Screening Visit 1 or planned during the coming year.

   General medical history
10. Weight <40 kg at Screening Visit 2.
11. Current smoking within the 12 months prior to Screening Visit 1 or a smoking history of >10 pack-years. Smoking includes tobacco, vaping, and/or marijuana use.
12. Known or suspected alcohol or drug abuse
13. Uncontrolled severe hypertension: systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg prior to the Baseline Visit despite antihypertensive therapy.
14. History of malignancy that required surgery (excluding local and wide-local excision), radiation therapy and/or systemic therapy during the 5 years prior to the Baseline Visit.
15. History of human immunodeficiency virus (HIV) infection or chronic infection with hepatitis B or C.
16. A helminth parasitic infection diagnosed within 24 weeks prior to Screening Visit 1 that has not been treated with or has failed to respond to standard of care (SoC) therapy.
17. Medical or other condition likely to interfere with participant's ability to undergo study procedures, adhere to visit schedule, or comply with study requirements.
18. Known or suspected noncompliance with medication.
19. Unwillingness or inability to follow the procedures outlined in the protocol.

    Clinical safety labs
20. Absolute neutrophil count (ANC) <2.000x10⁹/L at Screening Visit 1 or Screening Visit 2.
21. Renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m² at Screening Visit 2 (using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula for age ≥18 years at screening; using the Bedside Schwartz eGFR formula).
22. Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or unexplained elevations in alanine aminotransferase (ALT), aspartate aminotransferase (AST), >3x the upper limit of normal (ULN), or total bilirubin >2x ULN at Screening Visit 2 confirmed by a repeat abnormal measurement of the relevant value(s), at least 1 week apart.

    Cardiac safety
23. History of New York Heart Association class IV heart failure or last known left ventricular ejection fraction <25%.
24. History of major adverse cardiovascular event (MACE) within 3 months prior to the Baseline Visit.
25. History of cardiac arrhythmia within 3 months prior to the Baseline Visit that is not controlled by medication or via ablation.
26. History of long QT syndrome.
27. Corrected QT interval by Fridericia (QTcF) interval >450 ms for males and >470 ms for females at Screening Visit 2 or QTcF ≥480 ms for participants with bundle branch block.
28. Clinically important abnormalities in resting ECG that may interfere with the interpretation of QTcF interval changes at Screening Visit 2, including heart rate <45 beats per minute (bpm) or >100 bpm.

    Pregnancy/Lactation
29. Pregnant women or women breastfeeding
30. Males who are unwilling to use an acceptable method of birth control during the entire study period (ie, condom with spermicide).

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1061 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Annualized rate of severe asthma exacerbations over 52 weeks. | Day 1 (baseline, pre-dose) through Week 52
  A severe exacerbation was defined as a deterioration of asthma requiring: use of systemic corticosteroids for >=3 days; or hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids; or death due to asthma.

SECONDARY OUTCOMES:
Absolute Change in pre-bronchodilator forced expiratory volume (Pre-BD FEV)₁ from Baseline | Day 1 (baseline, pre-dose), Weeks 36, 44, 52
  The absolute change from baseline in pre-bronchodilator forced expiratory volume, averaged across visits at Weeks 36, 44, and 52.
Change From Baseline in Asthma Control Questionnaire-6 (ACQ-6) | Day 1 (baseline, pre-dose), Weeks 36, 44, 52
  Asthma Control Questionnaire-6 (ACQ-6), change from baseline, averaged across visits at Weeks 36, 44, and 52.
Change in Standardized version of the Asthma Quality of Life Questionnaire for 12 years and older (AQLQ+12) from baseline to Week 52. | Day 1 (baseline, pre-dose) through Week 52
Annualized rate of severe exacerbations requiring an emergency department visit or hospitalization over 52 weeks. | Day 1 (baseline, pre-dose) through Week 52
Annualized Rate of severe exacerbations from Week 4 to Week 52 | Week 4 through Week 52
Average change in absolute eosinophil count (AEC) | Day 1 (baseline, pre-dose) Weeks 36, 44, 52
Average change from baseline in forced vital capacity (FVC) | Day 1 (baseline, pre-dose), Weeks 36, 44, 52
Change from baseline in forced vital capacity (FVC) | Day 1 (baseline, pre-dose), Weeks 4, 12, 20,28 36, 44, 52
Change from baseline in Post-bronchodilator FEV₁ | Day 1 (baseline, pre-dose) through Week 52
Change from baseline in peak expiratory flow (PEF) | Day 1 (baseline, pre-dose) through Week 52
Time to first severe asthma exacerbation | Up to Week 52
Change from baseline in total asthma symptom score | Day 1 (baseline, pre-dose) through Week 52
Change from baseline in the EuroQol five-dimensional questionnaire (EQ-5D-5L) | Day 1 (baseline, pre-dose) through Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Salman Siddiqui, MD, Principal Investigator — Imperial College Healthcare NHS Trust (via Imperial Consultants)
Locations (400):
- United States (89):
  - Research Site 20001-374, Bakersfield, California
  - Research Site 20001-440, La Palma, California
  - Research Site 20001-062, Newport Beach, California
  - Research Site 20001-043, Newport Beach, California
  - Research Site 20001-380, Redding, California
  - Research Site US-20001-488, San Diego, California
  - Research Site 20001-003, West Covina, California
  - Research Site 20001-419, Westminster, California
  - Research Site 20001-048, Aventura, Florida
  - Research Site 20001-005, Brandon, Florida
  - Research Site 20001-051, Brandon, Florida
  - Research Site 20001-029, Coral Gables, Florida
  - Research Site 20001-350, Gainesville, Florida
  - Research Site 20001-014, Green Acres, Florida
  - Research Site 20001-054, Hialeah, Florida
  - Research Site 20001-067, Hialeah, Florida
  - Research Site 20001-020, Homestead, Florida
  - Research Site 20001-015, Kissimmee, Florida
  - Research Site 20001-002, Kissimmee, Florida
  - Research Site 20001-086, Loxahatchee Groves, Florida
  - Research Site 20001-066, Miami, Florida
  - Research Site 20001-001, Miami, Florida
  - Research Site 20001-059, Miami, Florida
  - Research Site 20001-026, Miami, Florida
  - Research Site 20001-065, Miami, Florida
  - Research Site 20001-024, Miami, Florida
  - Research Site 20001-069, St. Petersburg, Florida
  - Research Site 20001-004, Tampa, Florida
  - Research Site 20001-075, Augusta, Georgia
  - Research Site 20001-018, Columbus, Georgia
  - Research Site 20001-459, Sugar Hill, Georgia
  - Research Site 20001-090, Berwyn, Illinois
  - Research Site 20001-476, Chicago, Illinois
  - Research Site 20001-358, Normal, Illinois
  - Research Site 20001-135, River Forest, Illinois
  - Research Site 20001-403, Skokie, Illinois
  - Research Site 20001-036, Elwood, Indiana
  - Research Site 20001-044, Evansville, Indiana
  - Research Site 20001-021, Iowa City, Iowa
  - Research Site 20001-019, Owensboro, Kentucky
  - Research Site 20001-466, Baltimore, Maryland
  - Research Site 20001-456, Takoma Park, Maryland
  - Research Site 20001-055, White Marsh, Maryland
  - Research Site 20001-468, Fall River, Massachusetts
  - Research Site 20001-006, Flint, Michigan
  - Research Site 20001-148, Flint, Michigan
  - Research Site 20001-463, Rochester Hills, Michigan
  - Research Site 20001-370, Chesterfield, Missouri
  - Research Site 20001-074, Saint Charles, Missouri
  - Research Site 20001-046, St Louis, Missouri
  - Research Site 20001-409, Missoula, Montana
  - Research Site 20001-486, Henderson, Nevada
  - Research Site 20001-473, Las Vegas, Nevada
  - Research Site 20001-471, Highland Park, New Jersey
  - Research Site 20001-457, Jersey City, New Jersey
  - Research Site 20001-420, New Brunswick, New Jersey
  - Research Site 20001-050, East Amherst, New York
  - Research Site 20001-047, Hawthorne, New York
  - Research Site 20001-422, Rochester, New York
  - Research Site 20001-368, The Bronx, New York
  - Research Site 20001-408, Charlotte, North Carolina
  - Research Site 20001-039, Gastonia, North Carolina
  - Research Site 20001-435, Greenville, North Carolina
  - Research Site 20001-382, Raleigh, North Carolina
  - Research Site 20001-034, Cincinnati, Ohio
  - Research Site 20001-013, Cincinnati, Ohio
  - Research Site 20001-017, Dayton, Ohio
  - Research Site 20001-063, Toledo, Ohio
  - Research Site 20001-038, Edmond, Oklahoma
  - Research Site 20001-079, Oklahoma City, Oklahoma
  - Research Site 20001-395, Hershey, Pennsylvania
  - Research Site 20001-032, Columbia, South Carolina
  - Research Site 20001-025, Greenville, South Carolina
  - Research Site 20001-073, Spartanburg, South Carolina
  - Research Site 20001-438, Dickson, Tennessee
  - Research Site 20001-068, Amarillo, Texas
  - Research Site 20001-023, Dallas, Texas
  - Research Site 20001-028, Dallas, Texas
  - Research Site 20001-064, Houston, Texas
  - Research Site 20001-085, Houston, Texas
  - Research Site 20001-478, Plano, Texas
  - Research Site 20001-072, The Woodlands, Texas
  - Research Site 20001-258, Murray, Utah
  - Research Site 20001-477, Salt Lake City, Utah
  - Research Site 20001-340, Burke, Virginia
  - Research Site 20001-479, Vienna, Virginia
  - Research Site 20001-480, Barboursville, West Virginia
  - Research Site 20001-433, La Crosse, Wisconsin
  - Research Site 20001-057, Madison, Wisconsin
- Argentina (16):
  - Research Site 20054-054, Buenos Aires
  - Research Site -20054-021, Buenos Aires
  - Research Site 20054-023, Buenos Aires
  - Research Site 20054-011, Buenos Aires
  - Research Site 20054-017, Buenos Aires
  - Research Site 20054-015, Buenos Aires
  - Research Site 20054-022, Buenos Aires
  - Research Site 20054-024, Buenos Aires
  - Research Site 20054-008, Buenos Aires
  - Research Site 20054-005, Córdoba
  - Research Site 20054-019, Mendoza
  - Research Site 20054-016, Mendoza
  - Research Site 20054-010, Mendoza
  - Research Site 20054-013, Rosario
  - Research Site 20054-002, San Miguel de Tucumán
  - Research Site 20054-020, San Miguel de Tucumán
- Brazil (12):
  - Research Site 20055-012, Porto Alegre, Rio Grande do Sul
  - Research Site 20055-004, Porto Alegre, Rio Grande do Sul
  - Research Site 20055-014, Ribeirão Preto, São Paulo
  - Research Site 20055-009, Santos, São Paulo
  - Research Site 20055-001, São Bernardo do Campo, São Paulo
  - Research Site 20055-002, Sorocaba, São Paulo
  - Research Site 20055-007, Blumenau
  - Research Site 20055-011, Campo Largo
  - Research Site 20055-010, Porto Alegre
  - Research Site 20055-005, Santo André
  - Research Site 20055-003, São Paulo
  - Research Site 20055-008, São Paulo
- Bulgaria (22):
  - Research Site 20359-017, Dimitrovgrad
  - Research Site 20359-022, Kozloduy
  - Research Site 20359-027, Lovech
  - Research Site 20359-008, Montana
  - Research Site 20359-029, Montana
  - Research Site 20359-010, Pernik
  - Research Site 20359-023, Pleven
  - Research Site 20359-026, Plovdiv
  - Research Site 20359-024, Plovdiv
  - Research Site 20359-005, Rousse
  - Research Site 20359-009, Sliven
  - Research Site 20359-033, Sliven
  - Research Site 20359-025, Smolyan
  - Research Site 20359-014, Sofia
  - Research Site 20359-030, Sofia
  - Research Site 20359-020, Sofia
  - Research Site 20359-006, Sofia
  - Research Site 20359-015, Sofia
  - Research Site 20359-003, Stara Zagora
  - Research Site 20359-019, Stara Zagora
  - Research Site 20359-021, Velingrad
  - Research Site 20359-016, Vidin
- Canada (10):
  - Research Site 20011-011, Vancouver, British Columbia
  - Research Site 20011-019, Winnipeg, Manitoba
  - Research Site 20011-016, Ajax, Ontario
  - Research Site 20011-004, Ajax, Ontario
  - Research Site 20011-010, Burlington, Ontario
  - Research Site 20011-001, Windsor, Ontario
  - Research Site 20011-018, Montreal, Quebec
  - Research Site 20011-022, Québec, Quebec
  - Research Site 20011-020, Trois-Rivières, Quebec
  - Research Site 20011-024, Guelph
- China (37):
  - Research Site 20086-071, Jilin, Jilin
  - Research Site 20086-001, Taizhou, Zhejang
  - Research Site 20086-011, Baoding
  - Research Site 20086-037, Beijing
  - Research Site 20086-056, Beijing
  - Research Site 20086-012, Beijing
  - Research Site 20086-036, Beijing
  - Research Site 20086-057, Beijing
  - Research Site 20086-068, Beijing
  - Research Site 20086-002, Beijing
  - Research Site 20086-029, Beijing
  - Research Site 20086-076, Chengdu
  - Research Site 20086-072, Guandong
  - Research Site 20086-060, Guangdong
  - Research Site 20086-075, Guangxi
  - Research Site 20086-069, Guangzhou
  - Research Site 20086-039, Guizhou
  - Research Site 20086-050, Hangzhou
  - Research Site 20086-051, Hangzhou
  - Research Site 20086-059, Hangzhou
  - Research Site 20086-007, Hangzhou
  - Research Site 20086-022, Jinan
  - Research Site 20086-048, Luoyang
  - Research Site 20086-030, Nanchang
  - Research Site 20086-009, Nanchang
  - Research Site 20086-040, Ningbo
  - Research Site 20086-021, Pudong
  - Research Site 20086-019, Qingdao
  - Research Site 20086-061, Shanghai
  - Research Site 20086-063, Shanghai
  - Research Site 20086-052, Shanghai
  - Research Site 20086-041, Shanghai
  - Research Site 20086-053, Shenyang
  - Research Site 20086-064, Taiyuan
  - Research Site 20086-032, Weifang
  - Research Site 20086-066, Wuxi
  - Research Site 20086-017, Zhejiang
- Colombia (5):
  - Research Site 20057-008, Barranquilla
  - Research Site 20057-006, Bogotá
  - Research Site 20057-007, Ibagué
  - Research Site 20057-009, Santander
  - Research Site 20057-001, Zipaquirá
- Georgia (10):
  - Research Site 20995-007, Batumi
  - Research Site 20995-001, Kutaisi
  - Research Site 20995-005, Tbilisi
  - Research Site 20995-010, Tbilisi
  - Research Site 20995-006, Tbilisi
  - Research Site 20995-002, Tbilisi
  - Research Site 20995-003, Tbilisi
  - Research Site 20995-004, Tbilisi
  - Research Site 20995-009, Tbilisi
  - Research Site 20995-008, Tbilisi
- Japan (51):
  - Research Site 20081-080, Asahikawa
  - Research Site 20081-046, Fukuoka
  - Research Site 20081-003, Fukuoka
  - Research Site 20081-044, Fukuoka
  - Research Site 20081-025, Fukuoka
  - Research Site 20081-015, Gifu
  - Research Site 20081-077, Himeji
  - Research Site 20081-078, Hiroshima
  - Research Site 20081-071, Hokkaido
  - Research Site 20081-042, Ibaraki
  - Research Site 20081-069, Isehara
  - Research Site 20081-050, Kagoshima
  - Research Site 20081-079, Kobe
  - Research Site 20081-039, Kobe
  - Research Site 20081-072, Kochi
  - Research Site 20081-052, Kochi
  - Research Site 20081-090, Maebashi
  - Research Site 20081-030, Matsusaka
  - Research Site 20081-083, Miura
  - Research Site 20081-021, Nagoya
  - Research Site 20081-073, Nagoya
  - Research Site 20081-056, Niigata
  - Research Site 20081-037, Okayama
  - Research Site 20081-088, Ono
  - Research Site 20081-086, Osaka
  - Research Site 20081-024, Osaka
  - Research Site 20081-068, Osaka
  - Research Site 20081-041, Saga
  - Research Site 20081-076, Saitama
  - Research Site 20081-009, Shibuya-ku
  - Research Site 20081-032, Shimane
  - Research Site 20081-031, Shizuoka
  - Research Site 20081-061, Shizuoka
  - Research Site 20081-076, Tarumi
  - Research Site 20081-034, Tokyo
  - Research Site 20081-028, Tokyo
  - Research Site 20081-023, Tokyo
  - Research Site 20081-026, Tokyo
  - Research Site 20081-066, Tokyo
  - Research Site 20081-019, Tokyo
  - Research Site 20081-074, Tokyo
  - Research Site 20081-065, Tokyo
  - Research Site 20081-029, Tokyo
  - Research Site 20081-062, Toyama
  - Research Site 20081-038, Toyama
  - Research Site 20081-049, Tsuchiura
  - Research Site 20081-016, Yamaguchi
  - Research Site 20081-011, Yokohama
  - Research Site 20081-051, Yokohama
  - Research Site 20081-087, Yonago
  - Research Site 20081-043, Yoshida
- Lebanon (7):
  - Research Site 20961-007, Aïn Ouzaïn
  - Research Site 20961-003, Beirut
  - Research Site 20961-004, Beirut
  - Research Site 20961-009, Beirut
  - Research Site 20961-010, Beirut
  - Research Site 20961-012, Beirut
  - Research Site 20961-005, Tripoli
- Mexico (11):
  - Research Site 20052-011, Benito Juárez
  - Research Site 20052-008, Córdoba
  - Research Site 20052-035, Cuernavaca
  - Research Site 20052-002, Guadalajara
  - Research Site 20052-034, Guadalajara
  - Research Site 20052-013, Mérida
  - Research Site 20052-004, Mérida
  - Research Site 20052-012, San Juan del Río
  - Research Site 20052-037, San Nicolás de los Garza
  - Research Site 20052-006, Veracruz
  - Research Site 20052-009, Zapopan
- North Macedonia (6):
  - Research Site 20389-006, Shtip
  - Research Site 20389-003, Skopje
  - Research Site 20389-004, Skopje
  - Research Site 20389-007, Skopje
  - Research Site 20389-005, Strumica
  - Research Site 20389-001, Veles
- Peru (12):
  - Research Site 20051-009, Lima
  - Researcdh Site 20051-014, Lima
  - Research Site 20051-012, Lima
  - Research Site 20051-013, Lima
  - Research Site 20051-030, Lima
  - Research Site 20051-003, Lima
  - Research Site 20051-007, Lima
  - Research Site 20051-006, Lima
  - Research Site 20051-010, Lima
  - Research Site 20051-001, Lima
  - Research Site20051-002, Lima
  - Research Site 20051-008, Piura
- Poland (27):
  - Research Site 20048-001, Będzin
  - Research Site 20048-018, Bialystok
  - Research Site 20048-032, Bialystok
  - Research Site 20048-006, Giżycko
  - Research Site 20048-021, Katowice
  - Research Site 20048-002, Katowice
  - Research Site 20048-036, Kielce
  - Research Site 20048-027, Krakow
  - Research Site 20048-033, Krakow
  - Research Site 20048-008, Krakow
  - Research Site 20048-040, Krakow
  - Research Site 20048-005, Lodz
  - Research Site 20048-009, Lodz
  - Research Site 20048-015, Lodz
  - Research Site 20048-022, Lublin
  - Research Site 20048-024, Maków Podhalański
  - Research Site 20048-031, Ostrowiec Świętokrzyski
  - Research Site 20048-010, Piaseczno
  - Research Site 20048-028, Poznan
  - Research Site 20048-016, Poznan
  - Research Site 20048-039, Rzeszów
  - Research Site 20048-014, Skierniewice
  - Research Site 20048-037, Torun
  - Research Site 20048-012, Trzebnica
  - Research Site 20048-034, Warsaw
  - Research Site 20048-019, Wroclaw
  - Research Site 20048-029, Wroclaw
- Puerto Rico (2):
  - Research Site 20787-365, Guaynabo
  - Research Site 20787-390, Ponce
- Romania (6):
  - Research Site 20040-004, Brasov, Brașov County
  - Research Site 20040-006, Cluj-Napoca, Cluj
  - Research Site 20040-008, Bragadiru
  - Research Site 20040-002, Brasov
  - Research Site 20040-004, Brasov
  - Research Site 20040-011, Timișoara
- Serbia (12):
  - Research Site 20381-002, Belgrade
  - Research Site 20381-007, Belgrade
  - Research Site 20381-010, Belgrade
  - Research Site 20381-012, Belgrade
  - Research Site 20381-005, Belgrade
  - Research Site 20381-006, Belgrade
  - Research Site 20381-008, Kamenitz
  - Research Site 20381-001, Kragujevac
  - Research Site 20381-004, Niš
  - Research Site 20381-009, Novi Sad
  - Research Site 20381-011, Užice
  - Research Site 20381-003, Valjevo
- South Korea (12):
  - Research Site 20082-003, Anyang
  - Research Site 20082-007, Busan
  - Research Site 20082-009, Daegu
  - Research Site 20381-009, Incheon
  - Research Site 20082-006, Jeonju
  - Research Site 20082-013, Seoul
  - Research Site 20082-019, Seoul
  - Research Site 20082-008, Seoul
  - Research Site 20082-004, Seoul
  - Research Site 20082-014, Seoul
  - Research Site 20082-011, Seoul
  - Research Site 20082-010, Suwon
- Ukraine (21):
  - Research Site 20380-002, Chernivtsi
  - Research Site 20380-021, Chernivtsi
  - Research Site 20380-017, Ivano-Frankivsk
  - Research Site 20380-004, Ivano-Frankivsk
  - Research Site 20380-009, Ivano-Frankivsk
  - Research Site 20380-014, Ivano-Frankivsk
  - Research Site 20380-015, Kyiv
  - Research Site 20380-019, Kyiv
  - Research Site 20380-007, Kyiv
  - Research Site 20380-010, Kyiv
  - Research Site 20380-012, Kyiv
  - Research Site 20380-011, Kyiv
  - Research Site 20380-013, Kyiv
  - Research Site 20380-018, Kyiv
  - Research Site 20380-016, Lutsk
  - Research Site 20380-001, Ternopil
  - Research Site 20380-003, Vinnytsia
  - Research Site 20380-020, Vinnytsia
  - Research Site 20380-022, Vinnytsia
  - Research Site 20380-008, Vinnytsia
  - Research Site 20380-005, Zhytomyr
- United Kingdom (32):
  - Research Site 20044-001, Manchester, Greater Manchester
  - Research Site 20044-033, Manchester, Greater Manchester
  - Research Site 20044-046, Manchester, Greater Manchester
  - Research Site 20044-013, Manchester, Greater Manchester
  - Research Site 20044-008, Salford, Greater Manchester
  - Research Site 20044-010, Altrincham
  - Research Site 20044-079, Bedford
  - Research Site 20044-018, Bellshill
  - Research Site 20044-083, Birmingham
  - Research Site 20044-021, Birmingham
  - Research Site 20044-077, Bollington
  - Research Site 20044-017, Chorley
  - Research Site 20044-022, Enfield
  - Research Site 20044-019, Liverpool
  - Research Site 20044-084, London
  - Research Site 20044-081, London
  - Research Site 20044-036, London
  - Research Site 20044-042, London
  - Research Site 20044-020, Manchester
  - Research Site 20044-031, Manchester
  - Research Site 20044-032, Manchester
  - Research Site 20044-009, Manchester
  - Research Site 20044-005, Manchester
  - Research Site 20044-030, Manchester
  - Research Site 20044-012, Manchester
  - Research Site 20044-004, Manchester
  - Research Site 20044-082, Nottingham
  - Research Site 20044-024, Preston
  - Research Site 20044-026, Rochdale
  - Research Site 20044-029, Stockport
  - Research Site 20044-034, Stockport
  - Research Site 20044-078, Wythenshawe

IPD SHARING:
Plan to Share IPD: No